CLINICAL TRIAL: NCT01120990
Title: Validation of a Hybrid Blood Pressure Monitor to Replace the Mercury Standard for Validation Studies According to Modified Criteria of the European Society of Hypertension International Protocol 2010
Brief Title: Hybrid Blood Pressure Monitor Validation
Acronym: NISSEI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hybrid BP Monitor Validation
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Essential Hypertension
Keywords: Blood pressure measuring devices; Essential Hypertension; Automated blood pressure measurement
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Other): All eligible patients in the study consist a single group and the same intervention is assigned to all of them.
  Interventions: Other: Blood Pressure Measurement

INTERVENTIONS:
Other: Blood Pressure Measurement — All patients have their blood pressure measured simultaneously by two observers using parallel connected mercury sphygmomanometers and by a supervisor using the tested device, NISSEI DM 3000. Six sets of measurements are performed.

SUMMARY:
Assessment of the accuracy of a Blood Pressure Measuring Device with a digital display-column, NISSEI DM 3000, according to an adaptation of the "European Society of Hypertension International Protocol Revision 2010 for the Validation of Blood Pressure Measuring Devices in Adults".

DETAILED DESCRIPTION:
According to the "European Society of Hypertension International Protocol Revision 2010 for the Validation of Blood Pressure Measuring Devices in Adults", 33 patients have their blood pressure measured by two observers using parallel connected mercury sphygmomanometers, blinded from each other's result, and then by the supervisor using the tested device, NISSEI DM 3000. The measurements using the mercury sphygmomanometers are repeated 5 times and in between them, 4 measurements using the tested device take place. If the results of the comparison of these measurements according to the analysis required by the protocol, meet the required criteria, the device is regarded as "Pass", otherwise as "Fail".

In this study, instead of consecutive, simultaneous measurements of the two mercury sphygmomanometers and tha tested device will be taking place. This will be so to exclude any inaccuracy due to blood pressure variability and because the tested device has a controllable deflation rate and allows simultaneous measurements with the mercury sphygmomanometers. In addition, the investigators will be performing 6 set of measurements instead of 4.

ELIGIBILITY:
Inclusion Criteria:

* Above 25 years of age
* Sinus rhythm
* Informed consent

Exclusion Criteria:

* Sustained arrhythmia
* Pregnancy
* Poor quality Korotkoff sounds
* Unavailable cuff size
* Completed blood pressure range (according to protocol)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George S Stergiou, MD, Study Chair — Hypertension Center, Third Depertment of Medicine, University of Athens, Greece
Locations (1):
- Hypertension Center, Third Department of Medicine, University of Athens, Greece, Athens, Greece

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients included in the study with complete blood pressure measurements data consist a single group. The tested value is the degree of agreement between measurements performed with mercury devices and with the tested device
Period: Overall Study
Arm/Group | All Patients
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 50.4 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 31
Region of Enrollment [Number; unit: participants]
  Greece | 51

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Measured by Tested Device.
Description: Mean Systolic Blood pressure value of all BP measurements made by the tested device in all patients included in the analysis.
Time Frame: 3 months
Population: According to the European Society of Hypertension International Protocol 2010, recruitment is continued until 33 subjects that meet the entry criteria complete all the measurements.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 51
mmHg | 144.11 (27.72)

2. Primary Outcome: Systolic Blood Pressure Measured With Mercury Sphygmomanometer.
Description: Mean Systolic Blood pressure value of all BP measurements made by the two observers with mercury sphygmomanometers in all patients included in the analysis.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 51
mmHg | 143.92 (27.18)

3. Primary Outcome: Diastolic Blood Pressure Measured by Tested Device.
Description: Mean Diastolic Blood pressure value of all BP measurements made by the tested device in all patients included in the analysis.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 51
mmHg | 90.72 (20.02)

4. Primary Outcome: Diastolic Blood Pressure Measured With Mercury Sphygmomanometer.
Description: Mean Diastolic Blood pressure value of all BP measurements made by the two observers with mercury sphygmomanometers in all patients included in the analysis.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 51
mmHg | 90.51 (19.87)

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes